CLINICAL TRIAL: NCT07262996
Title: Comparison the Gender Effects of Knee Joint and Foot Complex Alignment During Single Leg Squat in Sedentaries
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: IstinyeUniversity
Record Dates: First submitted 2023-11-14; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-10

CONDITIONS: Woman's Role; Men's Role
Keywords: Single leg squat test; Q angle; Lower extremity alignment; Dynamic knee valgus; Navicular drop
MeSH Terms: interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men participants: Men participants between the ages of 18-30 years having an active lifestyle, able to squat without any pain or discomfort during the initial evaluation
  Interventions: Behavioral: Sociodemographic profile, dynamic valgus index, single leg squat test, Q angle, Foot posture index, navicular drop test, pain assessment, muscle strength and flexibility tests
- Women participants: Women participants between the ages of 18-30 years having an active lifestyle, able to squat without any pain or discomfort during the initial evaluation
  Interventions: Behavioral: Sociodemographic profile, dynamic valgus index, single leg squat test, Q angle, Foot posture index, navicular drop test, pain assessment, muscle strength and flexibility tests

INTERVENTIONS:
Behavioral: Sociodemographic profile, dynamic valgus index, single leg squat test, Q angle, Foot posture index, navicular drop test, pain assessment, muscle strength and flexibility tests — During the single leg squat test, they will be asked to perform a squat every two seconds without bending forward or sideways while maintaining their balance with their hands crossed over their chest. While performing the movement three (3) times in a slow and controlled manner, they will be recorded with a video camera positioned at 90 degrees to their full height (approximately 3m). This recording will be evaluated in computer environment with Kineovea 0.9.5 motion analysis program and dynamic valgus index will be calculated. Q angle will be measured with a goniometer in both standing and supine position. Medial longitudinal arch height will be measured by navicular drop test. Foot posture of the participants will be evaluated with the Foot Posture Index developed by Redmond et al. (2006) to evaluate foot posture.

SUMMARY:
In this study, the investigators aimed to investigate the relationship between the dynamic valgus index and the dynamic valgus index during the landing phase of the single leg squat movement of sedentary people according to gender and to evaluate the effect of the postural alignment of the ankle and foot complex on the stability of the knee joint during the single leg squat.

DETAILED DESCRIPTION:
Single leg squatting is the basis of many functional activities such as walking, running, landing and balance. Single leg squat is generally preferred for lower extremity rehabilitation and assessment of dynamic hip joint control, lower extremity kinematics and lower extremity alignment. Many studies have used single leg squats for knee kinematics assessment. Excessive knee valgus, hip adduction and abduction of the knee joint during the single leg squat pose a risk of injury to the anterior cruciate ligament, medial collateral ligament and other ligaments.

The single-leg squat test is frequently used clinically to provide a simple and convenient assessment of neuromuscular control for the lumbo-pelvic region. Misalignment of the lower limb can affect knee and hip kinematics during athletic movements, causing disorders such as anterior cruciate ligament lesions, iliotibial band syndrome and patellofemoral pain syndrome. The single leg squat test is a clinical functional test commonly used to assess clinical abnormal movement patterns of the lower limbs in terms of kinetic chain or coordinated muscle activity. This scale provides assessment of five dimensions: general impression, trunk posture, pelvis in space, hip joint movement and knee joint movement. Since the single-leg squat test tests both daily activity and lower limb balance ability during athletic tasks, it was deemed appropriate to perform it separately on both legs. It is a valid and reliable test preferred in the literature as a functional test that evaluates lower extremity and especially knee joint balance skills.

In the light of this information, the aim of this study was to investigate the relationship between the dynamic valgus index and the dynamic valgus index during the landing phase of the single leg squat movement of sedentary people according to gender and to evaluate the effect of the postural alignment of the ankle and foot complex on the stability of the knee joint during the single leg squat.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-30
* To have the physical capacity to perform single leg squat activity
* Voluntarily participate in the study

Exclusion Criteria:

* Current pain in the trunk and lower extremities
* Having a disease affecting the musculoskeletal system in the last six months
* History of surgery involving the lumbar region and lower extremities
* Having a neurological disease
* Having a disease that affects balance (such as vertigo)
* Diagnosis of a rheumatologic disease.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young adult persons
Study Population: Healthy young people who can perform the single leg squat activity
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Dynamic Valgus Index(DVI) | 3 months
  The mark between the participant's SIAS and the midpoint of the patella will be marked as the femur segment, and the mark between the patella and the foot will be marked as the tibia segment and video recording will be taken. Dynamic Valgus Index Measurement will be performed using Kineovea 0.9.5 motion analysis program. Knee frontal plane projection angle(KFPPA) will be measured with the computer program. The angle hip frontal plane projection angle(HFPPA) will be measured between the pelvis and the femur segment by determining the pelvis segment with the line connecting both SIAS marks. HFPPA will be subtracted from 90 degrees (90º - A) and KFPPA will be subtracted from 180 degrees (180º - B) and the DVI angle will be obtained by summing these two values.
Single leg squat test | 3 months
  The participants' spina iliaca anterior superior (SIAS) in the frontal plane, the middle of the patella on both sides, and the middle of the ankle will be marked by sticking red colored tape. The test protocol will be explained, visually demonstrated, and three (3) repetitions will be made to try and get used to the test. A T-shape will be drawn on the floor with tape to facilitate the evaluation and they will be asked to hold their free foot behind their back while standing barefoot. They will be asked to perform a squat every two seconds without leaning forward and sideways, while maintaining their balance with their hands crossed on their chest. While performing the movement three (3) times in a slow and controlled manner, they will be recorded with a video camera positioned at 90 degrees to their full height (approximately 3m). It will be observed on the video whether the participants are positioned in the straight midline towards the single leg squat test line. If the patella
Foot posture index | 3 months
  The participants' foot posture will be assessed using the Foot Posture Index developed by Redmond et al. (2006) to assess foot posture. It is mainly used to define the degree of supination, neutral or pronation position of the foot. All assessments are performed in a comfortable standing position with equal weight on both feet. This posture is reported to be close to the positions taken by the foot during the gait cycle. This index is composed of 6 assessment headings: palpation of the talus head, inclination above and below the lateral malleolus, calcaneal inversion/eversion assessment in the hindfoot, talonavicular alignment (concavity/convexity), medial arch height and forefoot abduction/adduction in the forefoot.
The demographic data of the participants | 3 months
  Age, gender, dominant limb, occupational status, working positions, sports practiced, if any, and weekly physical activity duration of the individuals included in the study will be recorded before the tests. The dominant limb will be determined as the limb preferred by the individuals for kicking the ball.
Weight of the participants | 3 months
  Weight of the participants were measured
Height of the participants | 3 months
  Height of the participants were measured
Body Mass Index(BMI) of the participants | 3 months
  BMI was calculated from weight and height data as kg/m^2

SECONDARY OUTCOMES:
Pain assessment | 3 months
  While performing the Squat Test, the participant will be asked if he/she has pain; if so, where it is located and will be asked to indicate the degree of pain with the Visual Analog Scale (VAS).
  Questions to be asked:
  Did you feel pain during squatting? If so, where did you feel pain? If you rate your pain on a visual scale (0 being the least and 10 being the most), how severe was the pain?

OTHER OUTCOMES:
Q angle | 3 months
  The anterosuperior iliac crista, midpoint of the patella and tibial tubercle will be marked while the person is in supine position. The Q-angle will be measured with a goniometer by intersecting a line drawn from the anterosuperior iliac crista to the midpoint of the patella and the proximal extension of a line drawn from the tibial tubercle to the midpoint of the patella. Q angle measurements will be repeated 3 times for each side lying and standing and averaged
Medial Longitudinal Arc Height | 3 months
  Medial Longitudinal Arch Height will be evaluated with the Navicular Drop Test. The height of the tubercle of the navicular bone above the ground will be recorded by marking on a white card while the participant is not transferring weight to the foot in a sitting position (A). Then, the height of the tubercle of the navicular bone above the ground will be marked while transferring equal weight to both feet in the standing upright position (B). The differences of the values taken during sitting and standing will be calculated and recorded in millimeters. Measurements will be taken for both sides and repeated 3 times and averaged
Tensor Fascia Lata Muscle Strength | 3 months
  Strength of the tensor fascia lata muscle will be assessed using standardized manual muscle testing procedures.
Quadriceps Muscle Strength | 3 months
  Strength of the quadriceps femoris muscle will be evaluated using manual muscle testing performed according to standardized clinical guidelines.
Hamstring Muscle Strength | 3 months
  Hamstring muscle strength will be measured using standardized manual muscle testing techniques.
Gastrocnemius-Soleus Muscle Strength | 3 months
  Strength of the gastrocnemius and soleus muscle group will be assessed using manual muscle testing with standardized patient positioning.
Tensor Fascia Lata Flexibility | 3 months
  Flexibility of the tensor fascia lata muscle will be assessed using the Modified Ober Test, and the hip adduction angle will be recorded.
Hamstring Flexibility | 3 months
  Hamstring flexibility will be evaluated using the Sit-and-Reach Test, and the maximal reach distance will be recorded.
Gastrocnemius Muscle Flexibility | 3 months
  The participant was positioned in supine, with the hip and knee placed in full extension. The knee to be tested was stabilized with one hand, while the examiner grasped the heel with the other hand and positioned their forearm along the plantar surface of the foot. The examiner then applied force to bring the foot into dorsiflexion. If the foot could not reach the neutral position (90°), the muscle was considered shortened.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap İnal, PhD, Study Director — Istanbul Galata University; Mehmet Onur Savaş, MSc.c, Principal Investigator — Istinye University
Locations (1):
- Gaziantep Şahinbey Ünaldı Aile Sağlığı Merkezi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gianola S, Castellini G, Stucovitz E, Nardo A, Banfi G. Single leg squat performance in physically and non-physically active individuals: a cross-sectional study. BMC Musculoskelet Disord. 2017 Jul 14;18(1):299. doi: 10.1186/s12891-017-1660-8. PMID 28709418
- [Background] Scholtes SA, Salsich GB. A DYNAMIC VALGUS INDEX THAT COMBINES HIP AND KNEE ANGLES: ASSESSMENT OF UTILITY IN FEMALES WITH PATELLOFEMORAL PAIN. Int J Sports Phys Ther. 2017 Jun;12(3):333-340. PMID 28593087
- [Background] Warner MB, Wilson DA, Herrington L, Dixon S, Power C, Jones R, Heller MO, Carden P, Lewis CL. A systematic review of the discriminating biomechanical parameters during the single leg squat. Phys Ther Sport. 2019 Mar;36:78-91. doi: 10.1016/j.ptsp.2019.01.007. Epub 2019 Jan 22. PMID 30703642